CLINICAL TRIAL: NCT06940648
Title: Virtuoso Improving Anatomic Bladder Lesion Excision Trial
Acronym: VIABLE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virtuoso Surgical, Inc. (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VES-173
Record Dates: First submitted 2025-04-04; First posted 2025-04-23 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Bladder Neoplasm
Keywords: Bladder Lesion; Resection; Excision; Bladder Tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Open label, single arm (Experimental): This study will enroll subjects 22 years and older with bladder lesions that require removal and/or biopsy for diagnosis, who meet all the inclusion criteria and none of the exclusion criteria. The study purpose is to evaluate the use of the Virtuoso Endoscopy System (VES) to perform safe and effective bladder lesion excisions.
  Interventions: Device: The study is to evaluate the use of the Virtuoso Endoscopy System to perform safe and effective bladder lesion excisions.

INTERVENTIONS:
Device: The study is to evaluate the use of the Virtuoso Endoscopy System to perform safe and effective bladder lesion excisions. — This study is to evaluate the use of the Virtuoso Endoscopy System (VES), which is a robotic enhanced system, to perform safe and effective bladder lesion excisions.

SUMMARY:
A robotic assisted surgery for bladder lesion excision.

DETAILED DESCRIPTION:
This is a single-center, non-randomized study to evaluate the use of the Virtuoso Endoscopy System (VES) to perform safe and effective bladder lesion excisions.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 22 years or older.
2. The subject is eligible and fit for transurethral bladder lesion removal and/or biopsy and has an appropriate indication to go through this surgery.
3. The subject is willing and able to provide written informed consent and comply with the study protocol.
4. The subject can undergo general anesthesia per anesthesiologist assessment.
5. The subject's aggregate bladder lesion(s) size is smaller than 3 cm.

Exclusion Criteria:

1. The subject has acute untreated urinary tract infection or urosepsis.
2. The subject has a documented nickel allergy or nickel sensitivity.
3. The subject is confirmed to be or suspected to be pregnant.
4. The subject is receiving anticoagulants and is unable or not willing to cease the medication for the investigational procedure.
5. The subject belongs to a vulnerable group (prisoner, etc.)
6. The subject has bladder dome or diverticular lesions that are at an increased risk for perforation of the bladder.
7. The subject's lesion(s) involve a ureteral orifice(s) necessitating additional endoscopic management and stenting.
8. The subject has a urethral abnormality, implant, or previous surgery which would conflict with the procedure.
9. The subject has undergone a transurethral bladder resection procedure in the past 6 months.
10. The subject has a history of radiation treatment within the pelvis.
11. Bladder tumor base maximal dimension is greater than 3 cm.
12. Bladder tumor detected during intravesical therapy.
13. Previous histological diagnosis different than non-muscle invasive bladder cancer.
14. Presence or prior history of upper urinary tract malignancy.
15. Eastern Cooperative Oncology Group performance status greater than or equal to 3.
16. American Society of Anesthesiologists physical status classification of III or above.
17. History of bleeding disorder, coagulation abnormality, or use of anticoagulants.
18. The presence of other active malignancy.
19. Life expectancy <1 yr.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Detrusor muscle presence in the pathologic specimen after VES procedure | Through study completion, an average of 30 days
Adverse events | Intraoperative
Adverse events | Through study completion, an average of 30 days

SECONDARY OUTCOMES:
Rate of conversion to standard cTURBT equipment | Intraoperative
Rate of en bloc or modified en bloc lesion excision with VES | Intraoperative
Complications (Clavien-Dindo) | Intraoperative
Significant bladder perforation requiring intervention | Intraoperative
Urethral injury | Intraoperative
Transfusion rate | Intraoperative
Estimated blood loss | Intraoperative
Rate of patients where the obturator nerve complex was observed | Intraoperative
Mortality | Intraoperative
VES surgery procedural time | Intraoperative
Presence of clear, evaluable margins in excised specimen | Through study completion, an average of 30 days
Time of catheterization | Through study completion, an average of 30 days
Time of hospital stay | Through study completion, an average of 30 days
Complications (Clavien-Dindo) | Through study completion, an average of 30 days
Significant bladder perforation requiring intervention | Through study completion, an average of 30 days
Urethral injury | Through study completion, an average of 30 days
30-day reoperation rate | Through study completion, an average of 30 days
30-day hospital readmission rate | Through study completion, an average of 30 days
30-day mortality | Through study completion, an average of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Teoh, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Teoh JY, Bracco FM, Wong JH, Liu AQ, Yuen VW, Lai FP. A Novel Transurethral Robotic Platform for Performing En Bloc Resection of Bladder Tumour: Results from the First Phase of the VIABLE Trial. Eur Urol Oncol. 2025 Nov 22:S2588-9311(25)00293-7. doi: 10.1016/j.euo.2025.11.005. Online ahead of print. PMID 41276423